CLINICAL TRIAL: NCT03837821
Title: A Window-of-opportunity Trial of Abemaciclib Followed by Radical Cystectomy in Patients With Platinum-ineligible Urothelial Carcinoma to Evaluate CDK4/6-dependent Phosphorylation of Pocket Proteins and Clonal Evolution Dynamics
Brief Title: (CLONEVO): Cell cycLe inhbitiON to Target the EVolution of UrOthelial Cancer
Acronym: CLONEVO
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1710018693
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): Abemaciclib 200 mg oral, every 12 hours
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib 200 mg oral, every 12 hours

SUMMARY:
Single-arm, open-label window-of-opportunity trial of neoadjuvant Abemaciclib in 20 patients, with tumor tissue obtained as standard of care at tumor resection (pre-Abemaciclib) and cystectomy (post-Abemaciclib)

DETAILED DESCRIPTION:
A Window-of-Opportunity Trial of Abemaciclib followed by radical cystectomy in patients with Platinum-Ineligible Urothelial Carcinoma to Evaluate CDK4/6-Dependent Phosphorylation of Pocket Proteins and Clonal Evolution Dynamics. Subjects will be treated with Abemaciclib at 200 mg every 12 hours for at least 4 weeks (and likely slightly longer depending upon surgical date). Individual dose reductions will be made on the basis of the AEs observed. In the absence of treatment delays due to adverse event(s), treatment will be continued until the surgical date unless any of the following criteria applies: 1-Disease progression; 2-Intercurrent illness that prevents further administration of treatment; 3-Unacceptable adverse event(s) as a result of Abemaciclib; 4- Patient decides to withdraw from the study; 5-General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator. Patients will be followed with history, physical, and blood tests at each visit to monitor for toxicity. Patients will be followed for survival endpoints following completion of this study for 3 years after surgery or until death. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years old at time of informed consent
2. Histologically confirmed MIBC (T2-T4) pure or mixed histology urothelial carcinoma [urothelial carcinoma should be the dominant (>50%) histology].
3. Refusing cisplatin-based chemotherapy or ineligible for cisplatin-based chemotherapy due to at least one of the following:

   1. Creatinine clearance < 60 mL/min (by Cockcroft-Gault calculation and/or measured creatinine clearance)
   2. Hearing loss ≥ grade 2 by CTCAE criteria and/or;
   3. Neuropathy ≥ grade 2 by CTCAE criteria and/or
   4. Heart failure NYHA ≥ III
4. Medically fit for TURBT and radical cystectomy
5. Adequate organ and marrow function as defined below:

   1. Absolute neutrophil count ≥ 1.5 K/mm3
   2. White blood cell count (WBC) > 3.0 K/mm3
   3. Platelets ≥ 100 K/mm3
   4. Hemoglobin ≥ 9 g/dL
   5. Serum total bilirubin ≤ 1.5 x ULN (Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted)
   6. ALT and AST ≤ 3.0 x ULN
6. Ability to swallow oral medications
7. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization

Exclusion Criteria

1. Patients with locally advanced unresectable or metastatic urothelial carcinoma as assessed on baseline radiographic imaging obtained within from the date of signed consent, 28 days prior to study enrollment. Low volume (<1.5 cm) suspicious lymph node metastases in the pelvis are allowed if they are in the LN dissection template field. The required radiographic imaging includes:

   1. Abdomen/pelvis - CT/MRI
   2. Chest - chest x-ray or CT scan
   3. Bone scan or FDG-PET/CT in the presence of bone pain or unexplained elevated alkaline phosphatase
2. Patients with another active second malignancy other than non-melanoma skin cancers and localized prostate cancer. Patients that have completed all necessary therapy and are considered to be <30% risk of relapse are not considered to have an active second malignancy and are eligible for enrollment.
3. Patients who have received anti-cancer therapy including chemotherapy, radiotherapy, immunotherapy, and monoclonal antibodies ≤ 4 weeks or 5 half-lives, whichever is longer, prior to starting study drug. Patients who received chemotherapy must have recovered to CTCAE Grade ≤1 from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to Cycle 1 Day 1. Patients currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor not to be scientifically or medically compatible with this study are also excluded.
4. Patients who have serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
5. Patients who have had major surgery within 14 days prior to Cycle 1 Day 1.
6. Have an active bacterial infection (especially if requiring IV antibiotics), systemic fungal and/or known viral infection (for example, human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C antibodies).
7. Subjects who received a strong CYP3A inhibitor within 7 days prior to the first dose of study drug, or patients who require continuous treatment with a strong CYP3A inhibitor
8. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
9. Pregnant or breast-feeding women
10. Women who do not agree to use a medically approved contraceptive method during the treatment period and for 3 weeks following the last dose of Abemaciclib
11. Men who do not agree to use a reliable method of birth control and to not donate sperm during the study and for at least 3 months following the last dose of Abemaciclib
12. Subjects unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in cell-cycle dynamics between pre- and post-Abemaciclib tumor samples | At baseline and post 4 week treatment
  Cell-cycle dynamics will be assessed by immunohistochemistry of tumor tissues, circulating tumor DNA (ctDNA) blood samples.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) of Abemaciclib | At baseline through 3 year follow up
  TEAEs will be assessed by utilizing the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Effect on tumor downstaging defined as <pT2 at time of cystectomy | At baseline and post 4 week treatment
  Tumor downstaging will be assess from tissue collected at the time of cystectomy.

OTHER OUTCOMES:
Impact of Abemaciclib on clonal evolution | Initiation of treatment up to 3 years
  Clonal evolution will be assessed by whole-exome sequencing and RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Bishoy Faltas, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Cornell Medicine, New York, New York
  - UT Southwestern Medical Center - Simmons Comprehensive Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No